CLINICAL TRIAL: NCT05150132
Title: The Effects of Interactive Powered Toothbrush With Application-assisted on Plaque, Gingivitis and Gingival Abrasion: A Randomized Controlled Clinical Trial.
Brief Title: Interactive Power Toothbrush With or Without App vs Manual Toothbrush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sühan Gürbüz, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2021-11-27; First posted 2021-12-08 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Toothbrushes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The examiner who performed clinical periodontal parameters was blinded to group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral-B Genius® 8000 power toothbrush with Cross Action brush head with smartphone app for 8 weeks (Experimental): Interactive PTB with Bluetooth® 4.0 connectivity smartphone app with Cross Action brush head using visually position detection feature. A triple pressure control system stops vibration, gives a visual warning, and reduces rotation speed in Daily Cleaning Mode-1.
  Interventions: Device: Oral-B Genius® 8000 power toothbrush with CrossAction brush head with smartphone app(Procter&Gamble,Ohio, USA)
- Oral-B Genius® 8000 power toothbrush with CrossAction brush head without smartphone app for 8 weeks (Active Comparator): PTB without Bluetooth® 4.0 connectivity without smartphone app with Cross Action brush head without using visually position detection feature triple pressure control system stops vibration, provides visual warning and reduces rotation speed. The group was asked to use PTB with daily cleaning mode 1 and brush head, but without using the Bluetooth app (without using the position detection system).
  Interventions: Device: Oral-B Genius® 8000 power toothbrush with CrossAction brush head without smartphone app(Procter&Gamble,Ohio, USA)
- Manual toothbrush: Oral B ClinicLine Pro-FlexSoft (Procter&Gamble,Ohio, USA) for 8 weeks (Active Comparator): They were instructed to brush according to the Modified Bass technique.
  Interventions: Device: Oral B ClinicLine Pro-FlexSoft (Procter&Gamble,Ohio, USA)

INTERVENTIONS:
Device: Oral-B Genius® 8000 power toothbrush with CrossAction brush head with smartphone app(Procter&Gamble,Ohio, USA) — All the participants were asked to brush with fluoride toothpaste (Pro-Expert Professional Protection- Ipana, Gross-Gerau, Germany) with a pea-sized amount (0.25 g) of the toothbrushes, which were given oral and applied instructions for use, twice a day in the morning and evening. The installation and operation of the toothbrush application (app) on the smartphone was activated in the PTB with the app group
  Arms: Oral-B Genius® 8000 power toothbrush with Cross Action brush head with smartphone app for 8 weeks
Device: Oral-B Genius® 8000 power toothbrush with CrossAction brush head without smartphone app(Procter&Gamble,Ohio, USA) — All the participants were asked to brush with fluoride toothpaste (Pro-Expert Professional Protection- Ipana, Gross-Gerau, Germany) with a pea-sized amount (0.25 g) of the toothbrushes, which were given oral and applied instructions for use, twice a day in the morning and evening. The installation and operation of the toothbrush application (app) on the smartphone were not activated in the PTB without the app group.
  Arms: Oral-B Genius® 8000 power toothbrush with CrossAction brush head without smartphone app for 8 weeks
Device: Oral B ClinicLine Pro-FlexSoft (Procter&Gamble,Ohio, USA) — All the participants were asked to brush with fluoride toothpaste (Pro-Expert Professional Protection- Ipana, Gross-Gerau, Germany) with a pea-sized amount (0.25 g) of the toothbrushes, which were given oral and applied instructions for use, twice a day in the morning and evening. They were instructed to brush with the Modified Bass technique.
  Arms: Manual toothbrush: Oral B ClinicLine Pro-FlexSoft (Procter&Gamble,Ohio, USA) for 8 weeks

SUMMARY:
It has been suggested that interactive power toothbrushes (PTBs), developed in recent years, provide more successful results in plaque control and effective use of brushing time by enabling patient collaboration and self-treatment, thanks to the application features associated with mobile phones. Interactive PTB synchronized with smartphones, including real-time feedback, session length, applications that prevent excessive brushing force, and focus brushing on specific areas with position detection technology, increases the brushing performance by increasing oral hygiene motivation.

Studies report that both power and manual toothbrushes cause gingival abrasion, a localized reversible lesion of the epithelium. While the opinions about the cause of gingival abrasion are not clear yet, the discussions regarding brush strength yet continue. While it is possible to control the interactive PTB force thanks to the mobile application, it is known that these high-speed rotating brushes control plaque effectively, but there is not enough evidence about its effect on gingival abrasion.

The primary purpose of this clinical study is to determine whether interactive PTB with application feature provides an additional benefit on plaque removal efficacy and reduction of gingival inflammation. In addition, this study aims to determine the effect of interactive power toothbrush with application on gingival abrasion by comparing it to interactive PTB without application and manual toothbrush. The study's null hypothesis in terms of gingival abrasion is that interactive PTB do not show a significant difference from other brushing methods.

ELIGIBILITY:
Inclusion Criteria:

* Dental students
* Diagnosed with gingivitis
* Clinical measurements: Probing pocket depths ≤3 mm, QHPI-TM ≥ 1.75 and with a bleeding site of at least 40% or more
* Aged between 18-25
* Non-smoker
* No systemic diseases
* Not undergoing orthodontic treatment
* No crowding
* No periodontal treatment in the last three months

Exclusion Criteria:

* Use of power toothbrush before
* Use of drugs that may affect the gingival tissues
* Having mucogingival problems
* Having carious teeth that require urgent treatment
* Probing pocket depths ˃ 3mm

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Turesky modification of the Quigley-Hein Plaque Index (QHPI-TM) index measurement | 2 weeks
  Tooth surfaces stained with Mira-2 Toneblue® were evaluated with six different scores: Score 0 = No plaque, Score 1 = Plaque stains on the cervical edge of the tooth, Score 2 = A thin, continuous strip of plaque (up to 1 mm) at the cervical edge of the tooth, Score 3 = band of plaque wider than 1 mm but covering less than one-third of the dental crown, Score 4 = Plaque covering at least one-third but less than two-thirds of the dental crown, Score 5 = Plaque covering two-thirds or more of the dental crown.
Turesky modification of the Quigley-Hein Plaque Index (QHPI-TM) index measurement | 8 weeks
  Tooth surfaces stained with Mira-2 Toneblue® were evaluated with six different scores: Score 0 = No plaque, Score 1 = Plaque stains on the cervical edge of the tooth, Score 2 = A thin, continuous strip of plaque (up to 1 mm) at the cervical edge of the tooth, Score 3 = band of plaque wider than 1 mm but covering less than one-third of the dental crown, Score 4 = Plaque covering at least one-third but less than two-thirds of the dental crown, Score 5 = Plaque covering two-thirds or more of the dental crown.
Bleeding on marginal bleeding index (BOMP) index measurement | 2 weeks
  The presence/absence and amount of bleeding were graded on a 0-2 scale within 30 seconds of probing by probing the gingival margin at an angle of approximately 60 to the long axis of the tooth (0 = no bleeding, 1 = punctate bleeding, 2 = excessive bleeding).
Bleeding on marginal bleeding index (BOMP) index measurement | 8 weeks
  The presence/absence and amount of bleeding were graded on a 0-2 scale within 30 seconds of probing by probing the gingival margin at an angle of approximately 60 to the long axis of the tooth (0 = no bleeding, 1 = punctate bleeding, 2 = excessive bleeding).
Staining with Mira-2 Toneblue® to detect the gingival abrasion scores | 2 weeks
  Blue or purple visible abrasions were classified by measuring with a Williams periodontal probe placed along the long axis of the lesions ("small" if ≤2 mm, "moderate" if ≥3 mm and ≤5 mm, and "large" if >5 mm).
Staining with Mira-2 Toneblue® to detect the gingival abrasion scores | 8 weeks
  Blue or purple visible abrasions were classified by measuring with a Williams periodontal probe placed along the long axis of the lesions ("small" if ≤2 mm, "moderate" if ≥3 mm and ≤5 mm, and "large" if >5 mm).

SECONDARY OUTCOMES:
Brushing times | 8 weeks
  The records in PTB group without-app and MTB were obtained with digital timer. In contrast, these records were obtained at the last appointment of the study; in Group PTB-A, the last brushing time records were sent to the researcher via e-mail by using the integral timer of the toothbrush, which is a feature of the mobile application.
Questionnaire | 8 weeks
  Questionnaire was applied to the participants including post-brushing pain/tenderness, cleaning capacity, manageability, and willingness to purchase via Visual Analogue Scale.
  Subjects were asked to mark a point on a 10 cm long uncalibrated line, with both ends interpreted as negative (left) or positive (right) ends.

CONTACTS AND LOCATIONS:
Locations (1):
- Sühan Gürbüz, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gurbuz S, Cankaya ZT, Cinal E, Kocyigit EG, Bodur A. Effects of interactive power toothbrush with or without application assistance on the plaque, gingivitis, and gingival abrasion among dental students: a randomized controlled clinical trial. Clin Oral Investig. 2022 Sep;26(9):5931-5941. doi: 10.1007/s00784-022-04553-3. Epub 2022 May 26. PMID 35614277